CLINICAL TRIAL: NCT06995131
Title: Evaluation of Aqueous Humor DEL-1 and IL-17 Levels in Diabetic Cataract Patients
Acronym: DEL-1 and IL-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Suzan Dogruya, Assistant professor, Uşak University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: DEL 1- IL 17
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Group (n=30); Non-diabetic Group
Keywords: Diabetes Mellitus; cataract; aqueous humor; Del 1; IL17
MeSH Terms: conditions — Diabetes Mellitus; Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: During the statistical analysis, the data analyst can analyze only "Group A" and "Group B" without knowing the group names. After the results are obtained, the groups are opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic cataract patients (Experimental): Collection of aqueous humor during cataract surgery in non-diabetic patients and study of DEL1 and IL 17
  Interventions: Diagnostic Test: Del 1; Diagnostic Test: IL 17
- Non-diabetic cataract patients (Sham Comparator): Collection of aqueous humor during cataract surgery in non-diabetic patients and study of DEL1 and IL 17
  Interventions: Diagnostic Test: Del 1; Diagnostic Test: IL 17

INTERVENTIONS:
Diagnostic Test: Del 1 — During cataract surgery, approximately 0.1-0.2 mL of aqueous humor will be sampled with a sterile 27 gauge syringe before viscoelastic is introduced into the anterior chamber. DEL 1 will be analyzed by ELISA
Diagnostic Test: IL 17 — During cataract surgery, approximately 0.1-0.2 mL of aqueous humor will be sampled with a sterile 27 gauge syringe before viscoelastic is introduced into the anterior chamber. IL 17 levels will be analyzed by ELISA

SUMMARY:
By comparing DEL-1 and IL-17 levels in the aqueous humor of diabetic cataract patients with the aqueous humor of non-diabetic patients, we aim to understand the biochemical effects of diabetes-related inflammatory processes in the eye.

DETAILED DESCRIPTION:
Developmental Endothelial Locus-1 (DEL-1) is a molecule related to endothelial cells and is a protein involved in intercellular interactions. It is generally associated with the development and function of endothelial cells lining the inner surface of the vessel. It plays an important role in the regulation of inflammation, the development of vessels and the organization of endothelial cells. It has also been shown to be associated with some types of cancer. It may also be effective in tissue regeneration and healing of injuries.

IL-17 (Interleukin-17) is a group of cytokines that play an important role in the immune system. There are several subtypes of IL-17, the best known and most researched being IL-17A. It regulates the body's immune response to certain infections. It is an important cytokine that initiates and supports the inflammation process. IL-17 plays an important role in the pathogenesis of various autoimmune and inflammatory diseases.

DEL-1 and IL-17 are two different molecules that act on inflammation and immune responses. DEL-1 helps regulate inflammation by protecting vascular health, while IL-17 can accelerate the course of diseases by increasing inflammation.

Diabetes is a systemic disease associated with oxidative stress and chronic inflammation. Retinopathy, cataract and glaucoma diseases develop due to diabetes. DEL-1 is a protein involved in the maintenance of vascular homeostasis and regulation of inflammation. Since diabetic patients have chronic inflammation and microvascular dysfunction, changes in DEL-1 levels may provide important clues to the pathophysiology

ELIGIBILITY:
Inclusion Criteria:

* Cataract diagnosed and surgery planned
* Patients without any other ocular pathology other than cataract.
* Type 2 DM for at least 5 years in the diabetic group

Exclusion Criteria:

* Patients with previous intraocular surgery
* Those with inflammatory eye diseases (e.g. uveitis)
* Those with autoimmune diseases or systemic inflammatory diseases
* Those receiving local or systemic steroid therapy
* Those with severe systemic disease (e.g. advanced renal failure, malignancy)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
DEL-1 and IL-17 levels | Perioperative
  To be measured quantitatively with ELISA kits, pg/mL

SECONDARY OUTCOMES:
Correlation between DEL-1 and IL-17 | Perioperative
  Pearson or Spearman correlation analyses will be used. pg/mL
Association of biomarker levels with HbA1c | Perioperative
  It will be analyzed by multivariate regression analysis.mmol/mol
Impact of demographic factors | Baseline
  The effect of age, gender and duration of diabetes on biomarkers will be statistically analyzed. Years, gender

CONTACTS AND LOCATIONS:
Locations (1):
- Uşak Training and Research Hospital, Uşak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) obtained in this study will be shared anonymised with requesting researchers for reasonable research purposes and in accordance with ethical rules.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The individual participant data (IPD) and related supporting information will be available starting 6 months after publication and will remain accessible for 5 years. Access will be granted to qualified researchers upon request, contingent on submission of an ethically approved research protocol.
Access Criteria: Researchers affiliated with academic institutions, clinicians, or independent scientists who provide an ethics committee-approved research protocol may request access.
URL: https://www.icmje.org/recommendations/browse/publishing-and-editorial-issues/clinical-trial-registration.html#fourth

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31076079/